CLINICAL TRIAL: NCT02052453
Title: ICD-ON Registry: Perioperative Management of Pacemakers and Implanted Cardioverter Defibrillators
Brief Title: ICD-ON Registry: Periop Management of Cardiac Devices
Status: Completed | Type: Observational
Sponsor: Edward Hospital (Other)
Collaborators: Medtronic (Industry); Abbott Medical Devices (Industry); Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Janet Gifford, Nurse Practitioner, Cardiology, Edward-Elmhurst Health System
Organization: Edward-Elmhurst Health System (Other)
Other Study IDs: ICDON2013
Record Dates: First submitted 2014-01-30; First posted 2014-02-03 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2016-07

CONDITIONS: Oversensing Cardiac Pacemaker; ICD; Surgery
Keywords: Pacemaker; ICD; Surgery; Electrocautery; Electromagnetic interference

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this registry is to document incidence of electrical magnetic interference (EMI), change in programmed parameters or device related events in patients with Pacemakers (PM) and Implanted Cardioverter Defibrillators (ICDs) having surgery requiring electrocautery. A standardized perioperative device management protocol (ICD-ON Protocol) will be used.

DETAILED DESCRIPTION:
Patients with PMs and ICDs have traditionally been considered at risk for electrical magnetic interference (EMI) from electrocautery. EMI can cause oversensing, pacing inhibition, or inappropriate ICD therapies. In July 2011, the Heart Rhythm Society /American Society of Anesthesiologists (HRS/ASA) published an Expert Consensus Statement on the perioperative management of PM and ICDs.

The purpose of this registry is to collect data on patients with PMs and ICDs undergoing procedures requiring electrocautery using a standardized device management protocol (ICD-ON Protocol). Decisions about management of patients with these devices will be made based on surgical location, programmed magnet response and pacemaker dependence.

This registry will document incidence of EMI, changes in programmed parameters or device related events associated with the procedures. Observational data will be collected on participants including: medical history, device parameters, surgical/cautery data, and postoperative device follow-up. For procedures not requiring reprogramming, postoperative PM and ICD interrogation will be either routine in office follow-up or remote monitoring, as per the subject's routine.

ELIGIBILITY:
* Have a implanted PM or ICD
* Be scheduled for a procedure with anticipated electrocautery
* Be able to speak, read and understand English
* Be willing to sign consent form

Exclusion Criteria:

* Have an ICD from Boston Scientific under Product Advisory related to magnet performance
* Have an ICD or PM from Biotronik or Sorin
* Surgical procedures with two or more electrocautery operators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have a PM or ICD undergoing procedures with anticipated electrocautery.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2014-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Incidence of EMI. | up to 90 days
  Percentage of patients with EMI, defined as oversensing on atrial or ventricular electrograms during electrocautery.

SECONDARY OUTCOMES:
Incidence of pacing inhibition in pacemaker dependent patients with procedures > 6 inches from device. | up to 90 days
  Percentage of patients with pacing inhibition recorded intraoperative or on postoperative electrograms during time of electrocautery.

OTHER OUTCOMES:
Incidence of device reset. | up to 90 days
  Percentage of total patients enrolled with device reset requiring reprogramming on their first postoperative interrogation. Either immediately postoperative for reprogramming group, in office or remote for all others.

CONTACTS AND LOCATIONS:
Overall Officials: Janet Gifford, MSN, NP, Principal Investigator — Edward Hospital
Locations (3):
- United States (3):
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Elmhurst Hospital, Elmhurst, Illinois
  - Edward Hospital, Naperville, Illinois

REFERENCES:
- [Background] Crossley GH, Poole JE, Rozner MA, Asirvatham SJ, Cheng A, Chung MK, Ferguson TB Jr, Gallagher JD, Gold MR, Hoyt RH, Irefin S, Kusumoto FM, Moorman LP, Thompson A. The Heart Rhythm Society (HRS)/American Society of Anesthesiologists (ASA) Expert Consensus Statement on the perioperative management of patients with implantable defibrillators, pacemakers and arrhythmia monitors: facilities and patient management this document was developed as a joint project with the American Society of Anesthesiologists (ASA), and in collaboration with the American Heart Association (AHA), and the Society of Thoracic Surgeons (STS). Heart Rhythm. 2011 Jul;8(7):1114-54. doi: 10.1016/j.hrthm.2010.12.023. No abstract available. PMID 21722856
- [Background] Gifford J, Larimer K, Thomas C, May P, Stanhope S, Gami A. Randomized controlled trial of perioperative ICD management: magnet application versus reprogramming. Pacing Clin Electrophysiol. 2014 Sep;37(9):1219-24. doi: 10.1111/pace.12417. Epub 2014 May 7. PMID 24802626